CLINICAL TRIAL: NCT04081909
Title: Opioid Free Anaesthesia vs Opioid Based Anesthesia in Cleft Lip, Palate ,Alveolus Surgery.
Brief Title: Opioid Based Anaesthesia vs Opioid Free Anesthesia in Cleft Lip, Palate ,Alveolus Surgery.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Yu Sun, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OFA vs OBA
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Intravenous Anesthesia
Keywords: Opioid; Ketamine; Dexmedetomidine; Sevoflurane; Perioperative complications
MeSH Terms: interventions — Ketamine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid Based Anesthesia(OBA) (Active Comparator)
  Interventions: Drug: Fentanyl，Remifentanil
- Opioid Free Anesthesia(OFA) (Experimental)
  Interventions: Drug: Ketamine,Dexmedetomidine

INTERVENTIONS:
Drug: Fentanyl，Remifentanil — Patients in OBA ,anesthesia induction will receive fentanyl 2ug/kg ,propofol 1% 2-3mg/kg, rocuronium 0.6-1mg/kg. Anesthesia maintenance with 1.5-2% sevoflurane, propofol 1% 3-6mg/kg/hr , remifentanil of 0.1- 0.2ug/ kg/ min.
  Arms: Opioid Based Anesthesia(OBA)
Drug: Ketamine,Dexmedetomidine — Patients in OFA,anesthesia induction will receive ketamine 1 mg/kg ,propofol 1% 2-3mg/kg, rocuronium 0.6-1mg/kg. Anesthesia maintenance with 1.5-2% sevoflurane, propofol 1% 3-6mg/kg/hr , dexmedetomidine of 0.4-0.8ug/ kg/ hr.
  Arms: Opioid Free Anesthesia(OFA)

SUMMARY:
Peri-operative opioid administration has long been one of the three pillars of 'balanced anaesthesia',over the span of just a few years,opioids were widely used in perioperative analgesia because of pain as the fifth vital sign.However, opioid administration is not without concern and is associated with many side-effects such as constipation, urinary retention, respiratory depression and postoperative nausea and vomiting .Cleft lip,palate,alveolus are common craniofacial abnormalities and usually require surgical repair.These patients have risks for various perioperative complications due to their young age and craniofacial abnormalities.

This study was designed to compare the effects of opioid based anesthesia（OBA） and opioid free anesthesia(OFA )on perioperative complications in patients with in cleft lip,palate,alveolus surgery, including respiratory depression, postoperative nausea and vomiting, hemodynamic effects, etc.

ELIGIBILITY:
Inclusion Criteria:

* American Society Anesthesia I, II；
* Age between 3 months and 12 years;

Exclusion Criteria:

* allergy to anesthetic and analgesic drugs;
* history of neuromuscular;
* renal, neurological, hepatic disease;
* cardiopulmonary diseases;
* bradycardia

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2019-09-04 (Estimated); Primary Completion 2020-05-04 (Estimated); Study Completion 2020-10-04 (Estimated)

PRIMARY OUTCOMES:
Respiratory depression | 24 hours following surgery
  Number of desaturation events (oxygen saturation by pulse oximetry (SPO2) <90%) during the first postoperative night's sleep

SECONDARY OUTCOMES:
Incidence of postoperative nausea and vomiting in the recovery room | first 2 postoperative hours
Incidence of postoperative nausea and vomiting on day 1 | 1st postoperative day
Severity of postoperative pain | 24 hours
  Comparison of the severity of postoperative pain in both group using the Face, Legs, Activity, Cry, Consolability scale for children between the ages of 3 months and 7 years. The scale has five criteria, which are each assigned a score of 0, 1 or 2.The scale is scored in a range of 0-10 with 0 representing no pain.
Severity of postoperative pain | 24 hours
  Comparison of the severity of postoperative pain in both group using Visual Analogue Scale for children aged 7 years and more. We instruct the patient to point to the position on the line between the faces to indicate how much pain they are currently feeling. The far left end indicates "no pain"(0) and the far right end indicates "worst pain ever."(10)
hemodynamic changes | Intraoperative
  blood pressure
hemodynamic changes | Intraoperative
  heart rate